CLINICAL TRIAL: NCT04841109
Title: Analysis of Diaphragm Movement During Its Postural Function Using M-mode Ultrasonography in Conjunction With Spirometry
Brief Title: Diaphragm Movement During Its Postural Function
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Martin Sembera, Clinical Professor, University Hospital, Motol
Other Study IDs: EK-237/21
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diaphragm Movement
Keywords: diaphragmatic motion; m-mode ultrasonography; postural function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to describe the movement of the diaphragm during postural activation of the trunk muscles in comparison with tidal breathing.

DETAILED DESCRIPTION:
Diaphragm movement will be measured by m-mode ultrasonography in a standing position. 30-35 healthy subjects will participate in the study. The movement of the diaphragm will be measured during tidal breathing then, during holding a load corresponding to 20% of the subject´s body weight and finally, during voluntary contraction of the trunk muscles. Trunk muscles contraction will be measured by a special device with pressure sensors placed on a trunk surface. Breathing activity will be measured by spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Able to comply with the study protocol, in the investigator's judgment
* Aged 20-40 years, inclusive
* Healthy as determined by the Investigator based on medical history, physical examination, vital signs and neurological examination
* Waist-to-height ratio < 0,59

Exclusion Criteria:

* Low back pain (acute or chronic)
* Previous abdominal or spine surgery
* Acute or chronic respiratory or musculoskeletal disorder
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks before initiation of the study
* Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Diaphragm movement | 6 months
  Distance of the diaphragm from the ultrasound transducer in millimeters during tidal breathing, during holding a load, and during voluntary contraction of the trunk muscles

SECONDARY OUTCOMES:
Tidal volume | 6 months
  Tidal volume in litres measured by spirometry during tidal breathing, during holding a load, and during voluntary contraction of the trunk muscles
Activity of the trunk muscles | 6 months
  Relative pressure in kilopascals generated by the trunk muscles during tidal breathing, during holding a load, and during voluntary contraction of these muscles

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kolar, Prof, PhD, Study Chair — Department of Rehabilitation and Sports Medicine, University Hospital Motol, Prague, Czech Republic
Locations (1):
- Pavel Kolar´s Centre of Physical Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sembera M, Busch A, Kobesova A, Hanychova B, Sulc J, Kolar P. The effect of abdominal bracing on respiration during a lifting task: a cross-sectional study. BMC Sports Sci Med Rehabil. 2023 Sep 15;15(1):112. doi: 10.1186/s13102-023-00729-w. PMID 37715283